CLINICAL TRIAL: NCT00718536
Title: Clinical Trial Assessing Once Daily Raltegravir Administration (800 mg QD) in HIV-1-Infected Patients Receiving Unboosted Atazanavir (400 mg QD)- Based Antiretroviral Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RALqd-ATV
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Atazanavir; Raltegravir; once-daily; pharmacokinetics; HIV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Addition of raltegravir 800 mg QD to HAART
  Interventions: Drug: Addition of raltegravir 800 mg QD to HAART

INTERVENTIONS:
Drug: Addition of raltegravir 800 mg QD to HAART — Addition of raltegravir 800 mg QD to HAART
  Other Names: HAART+RAL

SUMMARY:
The co-administration of raltegravir with medicinal products that are knouwn to be potent UGT1A1 inhibitors, such as atazanavir, may increase plasma levels of raltegravir. So once daily raltegravir (800 mg QD), instead of twice a day (400 mg BID), could be an appropriate therapeutic option in HIV-infected patients also receiving atazanavir-containing antiretroviral regimens. In this study, pharmacokinetic data supporting this hypothesis are recovered.

DETAILED DESCRIPTION:
Treatment adherence is crucial for the effectiveness of antiretroviral therapy, and, in an attempt to promote treatment adherence by the patients, once daily (QD) regimens are preferred rather than twice daily (BID) regimens.

The dose of 400 mg BID of raltegravir has been recently licensed for the treatment of human immunodeficiency virus (HIV-1) infection in treatment-experienced adult patients.

Raltegravir is eliminated mainly by metabolism via uridine diphosphate glucuronyl transferase (UGT1A1)-mediated glucuronidation pathway. Thus, co-administration of raltegravir with medicinal products that are known to be potent UGT1A1 inhibitors, such as atazanavir, may increase plasma levels of raltegravir.

Based on these data, it could be hypothesized that once daily raltegravir (800 mg QD) could be an appropriate therapeutic option in HIV-infected patients also receiving atazanavir-containing antiretroviral regimens. However, pharmacokinetic data supporting this hypothesis are lacking.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years old with documented HIV-1 infection.
2. Patients on antiretroviral regimen that includes atazanavir 400mg QD for at least 4 weeks.
3. Complete virological suppression (<50 copies/mL) for at least 12 months.
4. Voluntary written informed consent.
5. Ability of compliance with visit schedule.

Exclusion Criteria:

1. AIDS defining condition within 4 weeks prior to the initiation of the study.
2. Concomitant treatment with ritonavir as well as with inducers (NNRTI, rifampin, carbamazepine, phenytoin, phenobarbital, valproic acid, etc) or inhibitors (probenecid, etc) of the uridine diphosphate glucuronyl transferase within 2 weeks before the screening visit.
3. Concomitant therapy with tenofovir.
4. History or suspected poor adherence to HAART.
5. History of drug allergy to raltegravir

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Raltegravir area under the curve (AUC) 24 hours and Cmin | Day 10

SECONDARY OUTCOMES:
Adverse events | Baseline (BL), Day 10
Adherence | BL, Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Clotet Bonaventura, MD,PhD, Principal Investigator — Lluita contra la Sida Foundation, HIV Unit
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain